CLINICAL TRIAL: NCT05178355
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Doses Study of the Safety, Tolerability, and Pharmacokinetics of KVD824 Followed by Crossover Food Effect Sub-study in Healthy Volunteers
Brief Title: A Single and Multiple Doses Safety, Tolerability, Pharmacokinetics and Food Effect Study of KVD824 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KVD824-101
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part A - KVD824 - 10 mg (Experimental): 6 participants were administered10 mg of KVD824 in capsule form (1 x 10 mg capsule) on one occasion on Day 1. 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part A - KVD824 - 20 mg (Experimental): 6 participants were administered 20mg of KVD824 in capsule form ( 2 x 10 mg capsules) on one occasion on Day 1. 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part A - KVD824 - 40 mg (Experimental): 6 participants were administered 40mg of KVD824 in capsule form (1 x 40 mg capsule) on one occasion on Day 1. 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part A - KVD824 - 80 mg (Experimental): 6 participants were administered 80mg of KVD824 in capsule form (2 x 40 mg capsules) on one occasion on Day 1. 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part A - KVD824 - 160mg (Experimental): 6 participants were administered 160mg of KVD824 in capsule form (1 x 160 mg capsule) on one occasion on Day 1. 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part A - KVD824 - 320 mg (Experimental): 6 participants were administered 320mg of KVD824 in capsule form (1 x 320 mg capsule) on one occasion on Day 1. 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part A - KVD824 - 640 mg (Experimental): 6 participants were administered 640 mg of KVD824 in capsule form (2 x 320 mg capsule) on one occasion on Day 1. 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part A - KVD824 - 1280 mg (Experimental): 6 participants were administered 1280 mg of KVD824 in capsule form (4 x 320 mg capsule) on one occasion on Day 1. 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part B - KVD824 - 80 mg Multi-Dose (Experimental): 6 participants were administered 80 mg of KVD824 in capsule form (2 x 40 mg capsules) in multiple doses over a period of 5 days (twice a day on Days 1-4 and once in morning of Day 5; the first dose on each day was administered fasted). 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part B - KVD824 - 160 mg Multi-Dose (Experimental): 6 participants were administered 160mg of KVD824 in capsule form (1 x 160 mg capsule) in multiple doses over a period of 5 days (twice a day on Days 1-4 and once in morning of Day 5; the first dose on each day was administered fasted). 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part B - KVD824 - 320 mg Multi-Dose (Experimental): 6 participants were administered 320mg of KVD824 in capsule form (1 x 320 mg capsule) in multiple doses over a period of 5 days (twice a day on Days 1-4 and once in morning of Day 5; the first dose on each day was administered fasted). 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part B - KVD824 - 640 mg Multi-Dose (Experimental): 6 participants were administered 640mg of KVD824 in capsule form (2 x 320 mg capsules) in multiple doses over a period of 5 days (twice a day on Days 1-4 and once in morning of Day 5; the first dose on each day was administered fasted). 2 participants received matching placebo.
  Interventions: Drug: KVD824; Drug: Placebo to KVD824
- Part C - KVD824 - 320 mg Fasted (Experimental): 12 participants were administered 320 mg of KVD824 in capsule form (1 x 320 mg capsule) on one occasion on Day 1 in a fasted state.
  Interventions: Drug: KVD824
- Part C - KVD824 - 320 mg High fat breakfast (Experimental): 12 participants were administered 320 mg of KVD824 in capsule form (1 x 320 mg capsule) on one occasion on Day 1 following consumption of a high fat breakfast.
  Interventions: Drug: KVD824

INTERVENTIONS:
Drug: KVD824 — Active
Drug: Placebo to KVD824 — Placebo
  Arms: Part A - KVD824 - 10 mg; Part A - KVD824 - 1280 mg; Part A - KVD824 - 160mg; Part A - KVD824 - 20 mg; Part A - KVD824 - 320 mg; Part A - KVD824 - 40 mg; Part A - KVD824 - 640 mg; Part A - KVD824 - 80 mg; Part B - KVD824 - 160 mg Multi-Dose; Part B - KVD824 - 320 mg Multi-Dose; Part B - KVD824 - 640 mg Multi-Dose; Part B - KVD824 - 80 mg Multi-Dose

SUMMARY:
This is a 3 part phase 1, randomized, double-blind, placebo-controlled, study of the safety, tolerability, and pharmacokinetics of KVD824 following administration of single and multiple ascending oral doses; followed by a crossover food effect sub-study in healthy male volunteers.

DETAILED DESCRIPTION:
Part A was a single-centre randomized, double blinded, placebo control to investigate the safety and tolerability of single ascending doses of KVD824 administered to healthy male volunteers.

Part B was a single centre, randomized, double blinded, placebo control to investigate the safety and tolerability of multiple ascending doses of KVD824 administered to healthy male volunteers.

Part C was a single-centre, open labelled to investigate the food effect.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 and 55 years of age.
* Healthy subjects as determined by past medical history and as judged by the Chief Investigator / deputy.
* Male subject willing to wear a condom and whose partner of child bearing potential uses a highly effective method of contraception (e.g. partner use of intrauterine device (IUD)) or an effective method of contraception, i.e., established method of contraception + condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of IMP. Men whose partners are already pregnant must continue to use a condom during the trial and for three months thereafter.
* Subject with a body mass index (BMI) of 18-32 kg/m2.
* Subject with no clinically significant history of previous allergy / sensitivity to KVD824 or any of the excipients contained within the Investigational Medicinal Product.
* Subject with no clinically significant abnormal serum biochemistry, haematology, clotting profiles, and urine examination values within 28 days before the first dose of Investigational Medicinal Product.
* Subject with a negative urinary drugs of abuse screen, determined within 28 days before the first dose of Investigational Medicinal Product (N.B. a positive result may be repeated at the Chief Investigator's discretion).
* Subject with negative human immunodeficiency virus (HIV) and hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
* Subject with no clinically significant abnormalities in 12-lead electrocardiogram (QTcF ≤ 430 ms and PR interval 120-220 ms) determined within 28 days before first dose of Investigational Medicinal Product.
* Subject with no clinically significant abnormalities in vital signs (supine systolic (≤140 mmHg) and diastolic blood pressure (≤ 90 mmHg), pulse (≤ 100 bpm), oral temperature (≤ 37.5°C)) determined within 28 days before first dose of Investigational Medicinal Product.
* Subjects must not donate sperm from first dose until at least 3 months after last dose of Investigational Medicinal Product.
* Subjects without any special food restrictions that would hinder ability to consume gelatin (Part A and Part B placebo), or the high fat breakfast provided during study Part C; such as vegetarian, lactose intolerance, vegan, low-fat, low sodium, etc.
* Subjects with no known allergy or sensitivity to lactose and/or any additional excipients contained in Investigational Medicinal Product.
* Subject must be available to complete the study (including all follow up visits).
* Subject must satisfy the Chief Investigator / deputy about their fitness to participate in the study.
* Subject must provide written informed consent to participate in the study.

Exclusion Criteria:

* A clinically significant history of gastrointestinal disorder likely to influence Investigational Medicinal Product absorption.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 28 days or 5 half-lives (which ever is longer) prior to the first dose of Investigational Medicinal Product, unless in the opinion of the Chief Investigator the medication will not interfere with the study procedures or compromise subject safety.
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
* Subjects with a history of clotting abnormalities.
* A clinically significant history of drug or alcohol abuse in the last 5 years.
* Users of nicotine products i.e., current smokers or ex-smokers who have smoked within the 6 months prior to dosing with the study medication or users of cigarette replacements (e.g., e-cigarettes, nicotine patches or gums).
* Inability to communicate well with Investigators (i.e., language problem, poor mental development or impaired cerebral function).
* Participation in a New Chemical Entity clinical study within the previous 3 months or a marketed drug clinical study within the 30 days before the first dose of Investigational Medicinal Product. (Washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
* Donation of 450 mL or more blood within the 3 months before the first dose of Investigational Medicinal Product.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Safety - Treatment Emergent Adverse Events | Part A Days 0-10; Part B Days 0-12
  Number of Subjects with Treatment Emergent Adverse Events
Safety - Vital signs | Part A: Days (-1)-10;Part B: Days (-1)-12
  Number of participants with clinically significant changes in vital signs
Safety - Laboratory Parameters | Part A: Days (-1)-10;Part B: Days (-1)-12
  Number of participants with clinically significant changes in laboratory assessments
Safety - ECG change in QTcF | Part A: Days (-1)-10; Part B: Days (-1)-12
  Number of subjects who had any increase in QTcF parameters.

SECONDARY OUTCOMES:
Pharmacokinetic - Maximum Concentration (Cmax) | Part A: Predose and up to 18 samples over a 48 hour period post dose; Part B: Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5; Part C: Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of Cmax in all cohorts of Part A, B and C.
Pharmacokinetic - Time to maximum concentration (Tmax) | Part A: Predose and up to 18 samples over a 48 hour period post dose; Part B: Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5; Part C: Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of Tmax for Part A, Part B and Part C
Pharmacokinetic - Terminal Elimination Rate Constant (Kel) | Part A: Predose and up to 18 samples over a 48 hour period post dose; Part B: Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5; Part C: Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of Kel in Part A, Part B and Part C
Pharmacokinetic - Terminal elimination half-life (t1/2) | Part A: Predose and up to 18 samples over a 48 hour period post dose; Part B: Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5; Part C: Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of t1/2 in Part A, Part B and Part C
Pharmacokinetic - Area under the concentration-time curve from time 0 to 24 hour post dose (AUC0-24) | Part A: Predose and up to 18 samples over a 48 hour period post dose; Part B: Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5; Part C: Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of AUC (0-24) in Part A, Part B and Part C
Pharmacokinetic - Area under the concentration-time curve from time 0 to last measurable time-point (AUC0-t) | Part A: Predose and up to 18 samples over a 48 hour period post dose; Part B: Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5; Part C: Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of AUC (0-t) in Part A and Part C
Pharmacokinetic - Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | Part A: Predose and up to 18 samples over a 48 hour period post dose; Part B: Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5; Part C: Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of AUC (0-inf) in Part A, Part B and Part C
Pharmacokinetic - Residual Area under the curve (AUC%extrap) | Part A: Predose and up to 18 samples over a 48 hour period post dose; Part B: Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5; Part C: Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of AUC%extrap in Part A, Part B and Part C
Pharmacokinetic - Apparent total body clearance (CL/F) | Part A: Predose and up to 18 samples over a 48 hour period post dose; Part B: Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5; Part C: Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of CL/F in Part A, Part B and Part C
Pharmacokinetic - Apparent Volume of Distribution (Vz/F) | Part A: Predose and up to 18 samples over a 48 hour period post dose; Part B: Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5; Part C: Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of Vz/F in Part A, Part B and Part C
Pharmacokinetic - Area under the curve from time of first dose to 12 h post-dose (AUC0-12) | Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5
  Evaluation of AUC0-12 in Part B
Pharmacokinetic - Area under the curve from time of second dose to 12 h post-dose (AUC12-24) | Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5
  Evaluation of AUC12-24 in Part B
Pharmacokinetic - Apparent total body clearance at steady state (CLss/F) | Pre-dose and up to 11 samples over a 24 hour period post morning dose, day 1 and 5
  Evaluation of Clss/F in Part B
Pharmacokinetic - Maximum Concentration (Cmax) - Bioavailability Ratio Fed/Fasted | Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of Cmax Bioavailability Ratio Fed/Fasted in Part C
Pharmacokinetic - Area under the curve from the time of dosing to the time of the last measurable concentration (AUC 0-t) - Bioavailability Fed/Fasted Ratio | Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of AUC0-t Bioavailability Ratio Fed/Fasted in Part C
Pharmacokinetic - Area under the concentration-time curve from time 0 to infinity(AUC0-inf) - Bioavailability Fed/Fasted Ratio | Predose and up to 16 samples over a 24 hour period post dose per treatment period.
  Evaluation of AUC0-inf Bioavailability Ratio Fed/Fasted in Part C

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — KalVista Pharmaceuticals
Locations (1):
- KalVista Investigative Site, Merthyr Tydfil, United Kingdom